CLINICAL TRIAL: NCT05374408
Title: IDeA-CTR-Using Mobile Technology to Address the Trauma Mental Health Treatment Gap in Primary Care: Developing Implementation Protocols for Primary Care
Brief Title: Using Mobile Technology to Address the Trauma Mental Health Treatment Gap
Status: Completed | Type: Observational
Sponsor: University of Nebraska (Other)
Responsible Party: Sponsor
Other Study IDs: 0178-21-EP
Record Dates: First submitted 2022-05-03; First posted 2022-05-16 (Actual); Results first posted 2025-09-09 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-06

CONDITIONS: Post Traumatic Stress Disorder
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- BounceBack Now (BBN) Participants Aim 1: Participants who are receiving care at one of the designated integrated care clinics.
  Interventions: Behavioral: Aim 1 Participant Focus Groups
- BounceBack Now (BBN) Behavioral Health Provider Aim 1: Behavioral Health Providers who serve as a BHP at one of the designated integrated care clinics.
  Interventions: Behavioral: Aim 1 BHP Focus Groups
- BounceBack Now (BBN) Participants Aim 2: Participants who are receiving care at a designated integrated care clinic
  Interventions: Behavioral: Aim 2: BounceBack Now (BBN) for Trauma Informed Care Deployment; Behavioral: Aim 2 : Participant Focus Group
- Bounce Back Now (BBN) Aim 2 BHPs, Clinical Staff, Providers, and Administration: Clinical staff, Behavioral Health Providers, Providers, and Administration staff who can provide feedback pertaining to the factors that contribute to app deployment in an integrated care setting.
  Interventions: Behavioral: Aim 2: BHP, Provider, Staff and Admin Focus Groups

INTERVENTIONS:
Behavioral: Aim 2: BounceBack Now (BBN) for Trauma Informed Care Deployment — Brief explanation of BounceBack Now (BBN) will be provided. Participants will be directed to areas of the application that are congruent with treatment focus identified during their standard of care appointment.
  Participants will complete a baseline survey by either going online or being contacted by a member of the investigational team. The investigative assistant will contact all participants in 2-3 days to help the participant navigate the BBN and complete the baseline survey, if needed.
  The participant will continue to meet with their behavioral health provider (BHP) as determined by the standard of care interactions. BHP will highlight features contained in BBN for participant to use in between appointments.
  Follow-up phone calls will be scheduled for 2 weeks and 6 weeks after initial visit. During these phone- calls the participant will be contacted by a member of the investigational team to complete follow-up surveys.
  Groups: BounceBack Now (BBN) Participants Aim 2
Behavioral: Aim 1 Participant Focus Groups — At the beginning of the focus group the patients will be asked to download BBN on their smartphone device with the assistance of the research team, if they have not already done so. A basic tutorial of the BBN and the developed educational materials will be conducted/reviewed with the participants.
  After the tutorial and education has been provided the participants will be asked to try some of major features of the app. Then, they will be asked to review the patient education materials. They will be asked to discuss strengths and weaknesses of the materials. They will be also asked whether there is any content missing from the education material.
  Groups: BounceBack Now (BBN) Participants Aim 1
Behavioral: Aim 1 BHP Focus Groups — At the beginning of the focus group the BHPs will be asked to download BBN on their smartphone device with the assistance of the research team, if they have not already done so. A basic tutorial of the BBN and the developed educational materials will be conducted/reviewed with the BHPs.
  After the tutorial and education has been provided the participants will be asked to try some of major features of the app. Then, they will be asked to review the patient education materials. They will be asked to discuss strengths and weaknesses of the materials. They will be also asked whether there is any content missing from the education material.
  Groups: BounceBack Now (BBN) Behavioral Health Provider Aim 1
Behavioral: Aim 2: BHP, Provider, Staff and Admin Focus Groups — Semi-structured interviews will be conducted with BHPs, Clinical Staff, Providers and Administration They will ask questions to BHPs, Clinical Staff, Providers and Administration about feasibility, acceptability, and usability of BBN and overall clinical protocol.
  Groups: Bounce Back Now (BBN) Aim 2 BHPs, Clinical Staff, Providers, and Administration
Behavioral: Aim 2 : Participant Focus Group — Semi-structured interviews will be conducted with Participants to assess the feasibility, acceptability, and usability of BBN.
  Groups: BounceBack Now (BBN) Participants Aim 2

SUMMARY:
BounceBack Now (BBN) is a self-help, trauma-focused mental health mobile application (app) with automated assessment with treatment guidance and in-app evidence-based treatment support for depression, post-traumatic stress disorder (PTSD), sleep difficulties, and anxiety. BBN contains many of the necessary components to promote self-management of these conditions. Investigators will evaluate the app's feasibility and acceptability among under served participants (e.g., African Americans and participants with lower socioeconomic status) with trauma histories in an integrated primary care (IPC) setting. There are two specific aims: 1) to develop educational materials for patients and behavioral health providers for BBN in IPC, and 2) to conduct a pilot trial of BBN for participants with trauma histories in an IPC setting. For Aim 1, focus groups with behavioral health providers and participants will be conducted to obtain feedback about BBN and training materials. For Aim 2, a feasibility study with 15 participants will be conducted to identify and address any procedural issues and to refine the protocol before conducting the full-scale study.

DETAILED DESCRIPTION:
BounceBack Now (BBN) is a Trauma Focused Mobile Application. After consent, a behavioral health provider (BHP) will assist the participant in downloading BBN onto their smartphone device. The current BBN structure contains a brief assessment and multiple treatment components for disorders that are frequently associated with traumatic event exposure. A brief assessment based on the Kessler 6 will be completed and based on this assessment, the participants are then guided to treatment recommendations with an interactive rationale for each treatment. Education/explanations are provided in written, spoken, and animated video formats. Given that each of these treatments may be beneficial for patients with subsyndromal or very minor symptoms, all participants are able to see and interact with all treatment components, but it is anticipated that BHPs will provide recommendations for the sections that will be most beneficial. The treatment components are each based on effective in-person interventions. These include behavioral activation (depression), Written Exposure Therapy, and Expressive Writing (PTSD), Cognitive Behavioral Therapy for Sleep, and Relaxation/Mindfulness (stress/anxiety). The corresponding app sections are titled Activate, Write, Sleep, and Coping Tools, respectively. Each of these sections contains education components and there is a separate education component for the app overall that can be found through the coping tools page.

Aim 1: Develop educational materials for patients and Behavioral Health Providers (BHPs) for BBN in integrated primary care (IPC) settings. Investigators will present the educational materials and BBN in focus groups. These focus groups may be conducted virtually (i.e., zoom call) or in-person. The focus group will last 30 - 60 minutes. Focus groups will address acceptability, feasibility, and usability of the materials and the education materials and the app.

Focus groups will be audio recorded and a transcript will be prepared. Information obtained from the focus groups will be used to refine the patient and provider educational materials before we implement Aim 2 activities.

Aim 2: Conduct a pilot trial of BBN for participants with trauma histories in an IPC setting. A primary care provider at one of the two approved clinic locations will do a standard "warm handoff" referral to a behavioral health provider (BHP) if the patient is determined to have a behavioral health issue. The BHP will ask the patient about interest in participating the app study. If so, informed consent will be obtained and the participant screened using the Adverse Childhood Experience (ACE) screener to identify individuals at risk for trauma related conditions. Participants who screen positive on the ACE (>=3 points) will be invited to participate in further data collection for the study. A clinical assessment will be conducted, and a treatment assigned according to the standard of care specific to the mental health conditions of the participant. A brief explanation of BBN will be provided using the patient education material created under Aim 1. Certain features of the app will be suggested for use (e.g., journal, sleep intervention) according to participant need. The application is entirely self-paced, but a minimum use at least once a week is recommended.

Participants will complete a baseline survey online or through an investigational team member. Participants will continue to meet with their BHP as determined by the standard of care interactions, and, if deemed appropriate the BHP will highlight features contained in BBN for participant to use in between appointments. Follow-up phone calls will be scheduled for 2 week and 6 weeks after the initial visit to complete follow-up surveys, either online or administered by the investigative assistant over the phone. At the 6-week follow-up phone call, usability of the app will be assessed using the 18-item mHealth App Usability Questionnaire (MAUQ). Acceptability will be measured using the 20-item User Burden Scale. Additionally semi-structured interviews will be completed at that time or scheduled for an alternate date. The BHPs will complete a 5-item questionnaire about their comfort-level with integrating mental health apps into clinic care.

Addressing Needs of African American and Low-Income Patients:

The participating clinics primarily serve African American or low income patients. Race/ethnicity and income information will be collected through electronic health record data. The needs of these two patient population groups will be met by recruiting participants primarily from these two population groups for both aims to ensure their perspectives will be reflected in the patient education materials and by obtaining feedback through the individual interviews conducted at the end of the study.

ELIGIBILITY:
Inclusion Criteria:

Behavioral Health Providers:

• 19 years and older

Participants:

* 19 years and older
* Newly referred to a behavioral health provider at the Fontanelle or Midtown Clinic
* Own a smart phone

Exclusion Criteria

Behavioral Health Providers:

• 18 years and younger

Participants:

* 18 years and younger
* Referred to a behavioral health provider in the past year
* Does not own a smart phone
* Score 2 points or lower on the Adverse Childhood Experience screening
* High suicidality based on a clinical assessment by the behavioral health provider
* Having neurocognitive conditions either assessed by a primary care provider or diagnostic code for neurocognitive condition found in the patient note or Electronic Health Record (EHR)

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants with a trauma related disorder and behavioral health providers (BHPs) which are Clinical staff, providers and administration
Sampling Method: Non-Probability Sample
Enrollment: 29 (Actual)
Dates: Start 2022-08-03 (Actual); Primary Completion 2024-03-22 (Actual); Study Completion 2024-03-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Margaret R Emerson, DNP, APRN, Principal Investigator — University of Nebraska
Locations (2):
- United States (2):
  - Nebraska Medical Center-Fontenelle Clinic, Omaha, Nebraska
  - Nebraska Medical Center-Midtown Clinic, Omaha, Nebraska

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zhou L, Bao J, Setiawan IMA, Saptono A, Parmanto B. The mHealth App Usability Questionnaire (MAUQ): Development and Validation Study. JMIR Mhealth Uhealth. 2019 Apr 11;7(4):e11500. doi: 10.2196/11500. PMID 30973342
- [Background] Elwyn G, Frosch D, Thomson R, Joseph-Williams N, Lloyd A, Kinnersley P, Cording E, Tomson D, Dodd C, Rollnick S, Edwards A, Barry M. Shared decision making: a model for clinical practice. J Gen Intern Med. 2012 Oct;27(10):1361-7. doi: 10.1007/s11606-012-2077-6. Epub 2012 May 23. PMID 22618581
- [Background] Stetler CB, Damschroder LJ, Helfrich CD, Hagedorn HJ. A Guide for applying a revised version of the PARIHS framework for implementation. Implement Sci. 2011 Aug 30;6:99. doi: 10.1186/1748-5908-6-99. PMID 21878092

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: no pre-assignment details to report
Groups:
- Aim 1: Participant Focus Group: Participants who are receiving care at one of the designated integrated care clinics will participate in focus groups using semi-structured interviews to provide feedback about BBN along with educational materials to inform any changes needed prior to deployment of the app and education for Aim 2.
- Aim 1: Behavioral Health Provider Aim 1: semi-structured interviews will be conducted among BHPs at one of the designated clinics to review the educational materials prepared for BBN deployment.
- Aim 2: BounceBack Now (BBN) Participants: Deployment of BounceBack Now (BBN) for self-paced participant use
  BounceBack Now (BBN) for Trauma Informed Care: Brief explanation of BounceBack Now (BBN) will be provided. Participants will be directed to areas of the application that are congruent with treatment focus identified during their standard of care appointment.
  Participants will complete a baseline survey by either going online or being contacted by a member of the investigational team. The investigative assistant will contact all participants in 2-3 days to help the participant navigate the BBN and complete the baseline survey, if needed.
  The participant will continue to meet with their behavioral health provider (BHP) as determined by the standard of care interactions. BHP will highlight features contained in BBN for participant to use in between appointments.
  Follow-up phone calls will be scheduled for 2 weeks and 6 weeks after initial visit. During these phone- calls the participant will be contacted by a member of the investigational team to complete follow-up surveys.
- BHPS, Clinical Staff, Admin Aim 2: BHPS, Clinical Staff, Administrative Staff at one of the designated Integrated Care Clinic
Period: Overall Study
Arm/Group | Aim 1: Participant Focus Group | Aim 1: Behavioral Health Provider Aim 1 | Aim 2: BounceBack Now (BBN) Participants | BHPS, Clinical Staff, Admin Aim 2
Started | 5 | 2 | 12 | 10
Completed | 5 | 2 | 6 | 10
Not Completed | 0 | 0 | 6 | 0

BASELINE CHARACTERISTICS:
Population: Patients, BHPs, Clinical Staff, Providers and Administration individuals were recruited from designated integrated care clinical sites were recruited for Aim 1 and Aim 2 of the study.
Groups:
- Aim 1 BounceBack Now (BBN) Participants: Patients recruited to participate to in focus groups provide feedback about BBN and educational materials prior to app deployment..
- Aim 1 BounceBack Now (BBN) Behavioral Health Provider: BHPs were recruited to participate to in focus groups provide feedback about BBN and educational materials prior to app deployment
- Aim 2 BounceBack Now (BBN) Participants: Feasibility of integrating the BBN app into care
  BounceBack Now (BBN) for Trauma Informed Care: Brief explanation of BounceBack Now (BBN) will be provided. Participants will be directed to areas of the application that are congruent with treatment focus identified during their standard of care appointment.
  Participants will complete a baseline survey by either going online or being contacted by a member of the investigational team. The investigative assistant will contact all participants in 2-3 days to help the participant navigate the BBN and complete the baseline survey, if needed.
  The participant will continue to meet with their behavioral health provider (BHP) as determined by the standard of care interactions. BHP will highlight features contained in BBN for participant to use in between appointments.
  Follow-up phone calls will be scheduled for 2 weeks and 6 weeks after initial visit. During these phone- calls the participant will be contacted by a member of the investigational team to complete follow-up surveys.
- Aim 2 BounceBack Now (BBN) BHPs, Clinical Staff, Admin and Providers: BHPs, Clinical Staff, Admin and Providers were recruited to participate in focus groups to provide feedback about app use within the clinical setting.
- Total: Total of all reporting groups
Arm/Group | Aim 1 BounceBack Now (BBN) Participants | Aim 1 BounceBack Now (BBN) Behavioral Health Provider | Aim 2 BounceBack Now (BBN) Participants | Aim 2 BounceBack Now (BBN) BHPs, Clinical Staff, Admin and Providers | Total
Number analyzed (Participants) | 5 | 2 | 12 | 10 | 29
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 5 | 2 | 12 | 10 | 29
  >=65 years | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants] — Population: The gender was not collected for the BHP group
  Participants
    number analyzed (Participants) | 5 | 0 | 12 | 0 | 17
    Female | 3 |  | 11 |  | 14
    Male | 2 |  | 1 |  | 3
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: race was not collected for the BHPS
  Participants
    number analyzed (Participants) | 5 | 0 | 12 | 0 | 17
    American Indian or Alaska Native | 0 |  | 1 |  | 1
    Asian | 0 |  | 0 |  | 0
    Native Hawaiian or Other Pacific Islander | 0 |  | 0 |  | 0
    Black or African American | 2 |  | 2 |  | 4
    White | 3 |  | 6 |  | 9
    More than one race | 0 |  | 1 |  | 1
    Unknown or Not Reported | 0 |  | 2 |  | 2
Region of Enrollment [Number; unit: participants]
  United States | 5 | 2 | 12 | 10 | 29

OUTCOME MEASURES:

1. Primary Outcome: Aim 1: Evaluation of Educational Materials
Description: Educational Materials that have been developed related to using a trauma related mobile app will be evaluated by focus groups comprised of Patients and BHPs. The participants will be asked to use a think aloud approach using semi-structured interviews in order to determine the acceptability, usability and feasibility of the materials using questions developed to evaluate these items assessed during the focus group.
Time Frame: 5 months
Measure: Count of Participants; unit: Participants
Groups:
- BounceBack Now (BBN) Participants: Deployment of BounceBack Now (BBN) for self-paced participant use
  BounceBack Now (BBN) for Trauma Informed Care: Brief explanation of BounceBack Now (BBN) will be provided. Participants will be directed to areas of the application that are congruent with treatment focus identified during their standard of care appointment.
  Participants will complete a baseline survey by either going online or being contacted by a member of the investigational team. The investigative assistant will contact all participants in 2-3 days to help the participant navigate the BBN and complete the baseline survey, if needed.
  The participant will continue to meet with their behavioral health provider (BHP) as determined by the standard of care interactions. BHP will highlight features contained in BBN for participant to use in between appointments.
  Follow-up phone calls will be scheduled for 2 weeks and 6 weeks after initial visit. During these phone- calls the participant will be contacted by a member of the investigational team to complete follow-up surveys.
- BounceBack Now (BBN) Behavioral Health Provider: Feasibility of integrating the BBN app into care
  BounceBack Now (BBN) for Trauma Informed Care: Brief explanation of BounceBack Now (BBN) will be provided. Participants will be directed to areas of the application that are congruent with treatment focus identified during their standard of care appointment.
  Participants will complete a baseline survey by either going online or being contacted by a member of the investigational team. The investigative assistant will contact all participants in 2-3 days to help the participant navigate the BBN and complete the baseline survey, if needed.
  The participant will continue to meet with their behavioral health provider (BHP) as determined by the standard of care interactions. BHP will highlight features contained in BBN for participant to use in between appointments.
  Follow-up phone calls will be scheduled for 2 weeks and 6 weeks after initial visit. During these phone- calls the participant will be contacted by a member of the investigational team to complete follow-up surveys.
Arm/Group | BounceBack Now (BBN) Participants | BounceBack Now (BBN) Behavioral Health Provider
Number analyzed (Participants) | 5 | 2
Participants
  Acceptability | 3 | 2
  Usability | 4 | 2
  Feasibility | 3 | 2

2. Primary Outcome: Aim 2: Feasibility
Description: Feasibility will be assessed using semi-structured interviews. BHPs, Clinical Staff, Providers, Administration and Patients will complete semi-structured interviews guided by the Integrated Promoting Action on Research Implementation in Health Services Framework.
Time Frame: 8 months
Measure: Count of Participants; unit: Participants
Groups:
- BounceBack Now (BBN) Participants Focus Group: Participants who completed 6 weeks of the app use are asked to participate in semi-structured interviews to provide feedback on app use
- BounceBack Now BHP, Clinical Staff, Admin and Providers: Feasibility of integrating the BBN app into care focus group feedback
Arm/Group | BounceBack Now (BBN) Participants Focus Group | BounceBack Now BHP, Clinical Staff, Admin and Providers
Number analyzed (Participants) | 4 | 10
Participants
  Benefits of Use | 4 | 10
  Need for System Buy In | 2 | 7
  Systemic App Adoption Challenges | 2 | 8
  Implementation Challenges | 4 | 8
  Provider Specific Challenges | 1 | 10
  App Specific Adoption Challenges | 3 | 3

3. Primary Outcome: Aim 2: Acceptability: App Use
Description: Acceptability will also be measured by the number of patients who have downloaded and used the app for the duration of the 6 week study time-frame.
Time Frame: 8 months
Population: A total of 12 participants downloaded the app. N of 6 used the app for the duration of the study.
Measure: Count of Participants; unit: Participants
Arm/Group | BounceBack Now (BBN) Participants
Number analyzed (Participants) | 12
Participants | 6

4. Primary Outcome: Aim 2:Usability
Description: Patient usability of the app will be assessed using the 18-item mHealth App Usability Questionnaire (MAUQ). In this questionnaire each item is rated from 1 - strongly disagree, 2 - disagree, 3 - somewhat disagree, 4 - neither agree nor disagree, 5 - somewhat agree, 6 - agree, 7 - strongly agree. Scale Max= 126. Scale Min= 18
  To determine the usability of an app, calculate the total and determine the average of the responses to all of the 18 statements. The higher the overall average, the higher the usability of the app.
Time Frame: 8 months
Population: All participants (N=6) who completed the intervention and provided responses to the mHealth App Usability Questionnaire (MAUQ) at the post-intervention time point were included in the analysis. Responses marked as "Not Applicable" (NA) on individual items were excluded from the participant-level total score calculations. No participants were excluded from the analysis population.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | BounceBack Now (BBN) Participants
Number analyzed (Participants) | 6
score on a scale | 113.8 (6.7)

5. Primary Outcome: Aim 2: Patient Burden
Description: Patient acceptability, patients will complete the 20-item User Burden Scale at both follow-up visits. The scale has shown good overall inter-item reliability, convergent validity, and concurrent validity. The User Burden Scale (UBS) is a 20-item instrument used to assess perceived burden from digital health technologies across domains such as difficulty of use, time, physical demand, privacy, guilt, and financial burden. Each item is scored from 0 (Not at all) to 4 (Extremely), with total scores ranging from 0 (minimum) to 80 (Maximum). Higher scores indicate greater burden.
Time Frame: 8 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | BounceBack Now (BBN) Participants
Number analyzed (Participants) | 6
score on a scale | 4.17 (5.74)

ADVERSE EVENTS:
Time Frame: Adverse events data were collected through study completion, an average of 6 weeks per participant
Groups:
- BounceBack Now (BBN) Behavioral Health Provider Aim 1: BHPS who serve as a BHP at one of the designated integrated care clinics
- BounceBack Now Participants Aim 2: Participants who are receiving care at a designated integrated care clinic
- BounceBack Now Aim 2 BHPs, Clinical Staff, Providers, Admin: Clinical staff, BHPS, Providers and Admin staff who can provide feedback pertaining to factors that contribute to app deployment in the integrated setting.
Arm/Group | BounceBack Now (BBN) Participants Aim 1 | BounceBack Now (BBN) Behavioral Health Provider Aim 1 | BounceBack Now Participants Aim 2 | BounceBack Now Aim 2 BHPs, Clinical Staff, Providers, Admin
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/2 | 0/12 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/2 | 0/12 | 0/10
Other Adverse Events (participants affected / at risk) | 0/5 | 0/2 | 0/12 | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-02-28): https://cdn.clinicaltrials.gov/large-docs/08/NCT05374408/Prot_SAP_000.pdf